CLINICAL TRIAL: NCT01082055
Title: Retrospective Record Linkage Study to Investigate the Incidence of Complications and Follow-up Associated With Anti-arrythmic Drug Therapy
Brief Title: Antiarrythmic Drugs - Long-term Follow-up in the Modern Era
Status: Completed | Type: Observational
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Sponsor
Other Study IDs: ELD006
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2010-03

CONDITIONS: Cardiac Dysrhythmia
Keywords: Cardiac; Dysrhythmia; Safety
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Currently receiving antiarrythmic drugs

SUMMARY:
Antiarrhythmic drugs are associated with significant side effect profiles. Amiodarone has primarily class III action and whilst it has unrivalled efficacy in management of certain arrhythmias, it has a formidable side effect profile. Complications of continued therapy include, thyroiditis, hepatitis, cholestasis, increased skin sensitivity and pulmonary fibrosis. Current prescribing guidelines recommend frequent blood tests to monitor kidney, liver and thyroid function, in addition to frequent pulmonary function tests. Sotalol is a betablocker which possesses class III action in high doses and may predispose to QT prolongation Other class I agents such as flecainide and propafenone can be associated with sudden cardiac death in certain populations, and may predispose to other arrhythmias.

This study will examine the incidence of discontinuation of AAD therapy and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* At least one prescription for antiarrythmic drug

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients in Tayside receiving a prescription for an anti-arrythmic drug since 1994
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2010-03-01; Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Adverse Event | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Dundee, Dundee, United Kingdom